CLINICAL TRIAL: NCT00076011
Title: Phase 2 Study of AG 013736 as Second-Line Treatment in Patients With Metastatic Renal Cell Cancer
Brief Title: Anti-angiogenesis Agent AG-013736 in Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061012; NCT00077272 (obsolete NCT alias)
Record Dates: First submitted 2004-01-12; First posted 2004-01-14 (Estimated); Results first posted 2012-03-19 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms | interventions — Receptors, Vascular Endothelial Growth Factor; Receptors, Platelet-Derived Growth Factor

INTERVENTIONS:
Drug: Vascular Endothelial Growth Factor Receptor [VEGFR] and Platelet-Derived Growth Factor Receptor [PDGFR] inhibitor

SUMMARY:
The primary purpose of this protocol is to determine the activity of AG 013736 in patients with metastatic renal cell cancer who have received 1 prior cytokine-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented RCC with metastases.
* Failure of 1 prior cytokine-based therapy (interleukin-2 and/or interferon) due to disease progression or unacceptable treatment-related toxicity

Exclusion Criteria:

* Any prior systemic treatment for Renal Cell Carcinoma [RCC] other than 1 prior cytokine-based treatment regimen. Cytokine-based regimens containing thalidomide or an anti-angiogenesis agent are not allowed.
* Inability to take oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (6):
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Madison, Wisconsin
- Pfizer Investigational Site, Paris, Paris, France
- Pfizer Investigational Site, Hanover, Germany

REFERENCES:
- [Derived] Rixe O, Bukowski RM, Michaelson MD, Wilding G, Hudes GR, Bolte O, Motzer RJ, Bycott P, Liau KF, Freddo J, Trask PC, Kim S, Rini BI. Axitinib treatment in patients with cytokine-refractory metastatic renal-cell cancer: a phase II study. Lancet Oncol. 2007 Nov;8(11):975-84. doi: 10.1016/S1470-2045(07)70285-1. Epub 2007 Oct 23. PMID 17959415
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061012&StudyName=Anti-angiogenesis%20Agent%20AG-013736%20in%20Patients%20with%20Metastatic%20Renal%20Cell%20Carcinoma

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: Axitinib (AG-013736) tablet administered orally at a dose of 5 milligram (mg) twice daily (BID) in cycles of 4 weeks. Treatment was administered continuously until progression or unacceptable toxicity occurred.
Period: Overall Study
Arm/Group | Axitinib
Started | 52
Completed | 0
Not Completed | 52
Not completed — Death | 1
Not completed — Adverse Event | 10
Not completed — Lack of Efficacy | 25
Not completed — Withdrawal by Subject | 1
Not completed — Study terminated by sponsor | 3
Not completed — Other | 11
Not completed — Ongoing | 1

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 52
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non target). PR are those with at least 30 percent (%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline until the date of first documented progression or discontinuation from the study due to any cause, assessed every 8 weeks up to 139 weeks
Population: Study Population included all participants who received at least 1 dose of study medication and had a baseline assessment of disease.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 52
Percentage of participants | 44.2 [30.5 to 58.7]

2. Secondary Outcome: Time to Disease Progression (TTP)
Description: Time in days from start of study treatment to first documentation of objective tumor progression or death due to cancer, whichever comes first. TTP was calculated as (first event date minus the date of first dose of study medication plus 1). Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 52
Days | 477.0 [255.0 to 712.0]

3. Secondary Outcome: Duration of Response (DR)
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1). DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 1
Population: Subgroup of participants from the study population with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 23
Days | 700.0 [635.0 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to the high number of participants censored.

4. Secondary Outcome: Overall Survival (OS)
Description: Time in days from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1). Death was determined from adverse event (AE) data (where outcome was death) or from follow-up contact data (where the participant current status was death). For participants who were alive, overall survival was censored at the last contact.
Time Frame: Baseline to death due to any cause or at least 1 year after the initial dose for the last treated participant
Population: Study population included all participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 52
Days | 911.0 [619.0 to NA] — The upper limit of 95% CI was not estimable due to the high number of participants censored for survival.

5. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Version 3.0 (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms. Change from baseline=Cycle/Day score minus baseline score.
Time Frame: Baseline, Days 29, 57, 113, 169, 225, 281, 337, 393, 449, 505, 561, 617, 673, 729, 785, 841, 897, 953 and follow-up visit after last dose
Population: Study population included all participants who received at least 1 dose of study medication and had a baseline assessment of disease. The 'n' is signifying those participants who were evaluable for this measure at the specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Axitinib
Number analyzed (Participants) | 52
Units on a scale
  Global health status: Baseline (n=52) | 68.9 (23.05)
  Global health status: Change at Day 29 (n=46) | -6.0 (20.54)
  Global health status: Change at Day 57 (n=33) | -0.3 (24.60)
  Global health status: Change at Day 113 (n=41) | -4.9 (25.82)
  Global health status: Change at Day 169 (n=32) | -7.6 (28.58)
  Global health status: Change at Day 225 (n=28) | 4.8 (29.17)
  Global health status: Change at Day 281 (n=22) | 2.3 (24.42)
  Global health status: Change at Day 337 (n=14) | -0.6 (26.65)
  Global health status: Change at Day 393 (n=19) | 5.7 (24.85)
  Global health status: Change at Day 449 (n=16) | 6.3 (28.30)
  Global health status: Change at Day 505 (n=19) | 1.8 (30.75)
  Global health status: Change at Day 561 (n=16) | 2.6 (31.73)
  Global health status: Change at Day 617 (n=14) | -6.0 (34.35)
  Global health status: Change at Day 673 (n=11) | 5.3 (34.01)
  Global health status: Change at Day 729 (n=11) | 8.3 (28.87)
  Global health status: Change at Day 785 (n=10) | 9.2 (36.74)
  Global health status: Change at Day 841 (n=4) | -8.3 (29.66)
  Global health status: Change at Day 897 (n=1) | -16.7 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Global health status: Change at Day 953 (n=1) | -33.3 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Global health status: Change at follow-up (n=12) | -0.7 (17.57)
  Physical functioning: Baseline (n=52 ) | 80.6 (18.84)
  Physical functioning: Change at Day 29 (n=47) | -7.1 (16.08)
  Physical functioning: Change at Day 57 (n=45) | -2.6 (15.24)
  Physical functioning: Change at Day 113 (n=41) | -3.8 (15.38)
  Physical functioning: Change at Day 169 (n=32) | -5.9 (14.07)
  Physical functioning: Change at Day 225 (n=28) | -3.6 (17.11)
  Physical functioning: Change at Day 281 (n=23) | -2.7 (19.25)
  Physical functioning: Change at Day 337 (n=14) | -1.0 (18.09)
  Physical functioning: Change at Day 393 (n=19) | 1.8 (12.93)
  Physical functioning: Change at Day 449 (n=17) | -3.0 (18.45)
  Physical functioning: Change at Day 505 (n=20) | -3.0 (18.29)
  Physical functioning: Change at Day 561 (n=17) | -6.3 (21.79)
  Physical functioning: Change at Day 617 (n=14) | -3.8 (20.87)
  Physical functioning: Change at Day 673 (n=11) | 4.2 (15.57)
  Physical functioning: Change at Day 729 (n=11) | 4.2 (18.44)
  Physical functioning: Change at Day 785 (n=10) | -3.3 (19.18)
  Physical functioning: Change at Day 841 (n=5) | 6.7 (16.33)
  Physical functioning: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Physical functioning: Change at Day 953 (n=1) | -33.3 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Physical functioning: Change at follow-up (n=12) | -6.8 (17.53)
  Role functioning: Baseline (n=52 ) | 80.4 (26.55)
  Role functioning: Change at Day 29 (n=47) | -9.2 (28.62)
  Role functioning: Change at Day 57 (n=45) | -8.9 (22.64)
  Role functioning: Change at Day 113 (n=41) | -13.4 (32.32)
  Role functioning: Change at Day 169 (n=32) | -14.6 (25.66)
  Role functioning: Change at Day 225 (n=28) | -8.9 (31.26)
  Role functioning: Change at Day 281 (n=23) | -5.8 (23.36)
  Role functioning: Change at Day 337 (n=14) | -6.0 (19.18)
  Role functioning: Change at Day 393 (n=19) | -2.6 (23.08)
  Role functioning: Change at Day 449 (n=16) | -4.2 (34.69)
  Role functioning: Change at Day 505 (n=20) | -6.7 (29.32)
  Role functioning: Change at Day 561 (n=17) | -9.8 (32.84)
  Role functioning: Change at Day 617 (n=14) | -13.1 (32.14)
  Role functioning: Change at Day 673 (n=11) | -4.5 (27.98)
  Role functioning: Change at Day 729 (n=11) | 1.5 (31.14)
  Role functioning: Change at Day 785 (n=10) | -6.7 (32.58)
  Role functioning: Change at Day 841 (n=5) | 10.0 (27.89)
  Role functioning: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Role functioning: Change at Day 953 (n=1) | -33.3 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Role functioning: Change at follow-up (n=12) | -11.1 (22.84)
  Emotional functioning: Baseline (n=52) | 80.1 (19.40)
  Emotional functioning: Change at Day 29 (n=46) | -0.4 (19.22)
  Emotional functioning: Change at Day 57 (n=33) | 3.8 (16.55)
  Emotional functioning: Change at Day 113 (n=41) | -0.2 (15.08)
  Emotional functioning: Change at Day 169 (n=32) | -0.3 (16.86)
  Emotional functioning: Change at Day 225 (n=28) | 6.5 (22.26)
  Emotional functioning: Change at Day 281 (n=23) | 6.5 (17.40)
  Emotional functioning: Change at Day 337 (n=14) | 11.3 (19.78)
  Emotional functioning: Change at Day 393 (n=19) | 11.0 (17.36)
  Emotional functioning: Change at Day 449 (n=16) | 7.5 (23.69)
  Emotional functioning: Change at Day 505 (n=19) | 4.4 (21.04)
  Emotional functioning: Change at Day 561 (n=17) | 7.5 (21.17)
  Emotional functioning: Change at Day 617 (n=14) | 6.5 (21.23)
  Emotional functioning: Change at Day 673 (n=11) | 9.1 (24.28)
  Emotional functioning: Change at Day 729 (n=11) | 8.3 (25.82)
  Emotional functioning: Change at Day 785 (n=10) | 4.2 (20.13)
  Emotional functioning: Change at Day 841 (n=4) | 6.3 (21.92)
  Emotional functioning: Change at Day 897 (n=1) | 25.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Emotional functioning: Change at Day 953 (n=1) | -16.7 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Emotional functioning: Change at follow-up (n=12) | -3.5 (20.86)
  Cognitive Functioning: Baseline (n=52) | 86.5 (16.18)
  Cognitive Functioning: Change at Day 29 (n=46) | -2.5 (16.47)
  Cognitive Functioning: Change at Day 57 (n=33) | 1.0 (14.40)
  Cognitive Functioning: Change at Day 113 (n=41) | -5.3 (15.11)
  Cognitive Functioning: Change at Day 169 (n=32) | -7.8 (15.25)
  Cognitive Functioning: Change at Day 225 (n=28) | -6.5 (19.95)
  Cognitive Functioning: Change at Day 281 (n=23) | -2.2 (14.48)
  Cognitive Functioning: Change at Day 337 (n=14) | 0.0 (20.67)
  Cognitive Functioning: Change at Day 393 (n=19) | 0.9 (17.10)
  Cognitive Functioning: Change at Day 449 (n=16) | 0.0 (19.25)
  Cognitive Functioning: Change at Day 505 (n=19) | -0.9 (15.19)
  Cognitive Functioning: Change at Day 561 (n=17) | -1.0 (19.07)
  Cognitive Functioning: Change at Day 617 (n=14) | -4.8 (18.98)
  Cognitive Functioning: Change at Day 673 (n=11) | 1.5 (21.67)
  Cognitive Functioning: Change at Day 729 (n=11) | 3.0 (22.13)
  Cognitive Functioning: Change at Day 785 (n=10) | 0.0 (17.57)
  Cognitive Functioning: Change at Day 841 (n=4) | 0.0 (27.22)
  Cognitive Functioning: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Cognitive Functioning: Change at Day 953 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Cognitive Functioning: Change at follow-up (n=12) | -4.2 (16.09)
  Social functioning: Baseline (n=52) | 81.7 (26.46)
  Social functioning: Change at Day 29 (n=46) | -8.7 (29.97)
  Social functioning: Change at Day 57 (n=33) | -3.0 (31.31)
  Social functioning: Change at Day 113 (n=41) | -6.1 (27.07)
  Social functioning: Change at Day 169 (n=32) | -9.4 (31.09)
  Social functioning: Change at Day 225 (n=28) | -1.2 (38.74)
  Social functioning: Change at Day 281 (n=23) | 4.3 (28.08)
  Social functioning: Change at Day 337 (n=14) | -0.0 (35.20)
  Social functioning: Change at Day 393 (n=19) | 1.8 (26.58)
  Social functioning: Change at Day 449 (n=16) | -3.1 (30.56)
  Social functioning: Change at Day 505 (n=19) | -3.5 (35.82)
  Social functioning: Change at Day 561 (n=17) | -6.9 (33.88)
  Social functioning: Change at Day 617 (n=14) | -9.5 (32.50)
  Social functioning: Change at Day 673 (n=11) | 4.5 (35.03)
  Social functioning: Change at Day 729 (n=11) | 4.5 (36.58)
  Social functioning: Change at Day 785 (n=10) | 1.7 (36.39)
  Social functioning: Change at Day 841 (n=4) | 4.2 (20.97)
  Social functioning: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Social functioning: Change at Day 953 (n=1) | -66.7 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Social functioning: Change at follow-up (n=12) | -2.8 (23.39)
  Fatigue: Baseline (n=52) | 27.4 (23.64)
  Fatigue: Change at Day 29 (n=47) | 11.8 (24.54)
  Fatigue: Change at Day 57 (n=45) | 7.2 (22.27)
  Fatigue: Change at Day 113 (n=41) | 7.2 (22.58)
  Fatigue: Change at Day 169 (n=32) | 6.9 (18.24)
  Fatigue: Change at Day 225 (n=28) | 3.8 (28.37)
  Fatigue: Change at Day 281 (n=23) | 1.9 (24.31)
  Fatigue: Change at Day 337 (n=14) | 3.2 (24.82)
  Fatigue: Change at Day 393 (n=19) | -4.1 (22.59)
  Fatigue: Change at Day 449 (n=17) | -0.0 (26.64)
  Fatigue: Change at Day 505 (n=20) | 4.7 (25.44)
  Fatigue: Change at Day 561 (n=17) | 3.3 (26.28)
  Fatigue: Change at Day 617 (n=14) | 8.3 (24.92)
  Fatigue: Change at Day 673 (n=11) | -3.0 (25.38)
  Fatigue: Change at Day 729 (n=11) | -4.0 (27.79)
  Fatigue: Change at Day 785 (n=10) | -1.1 (30.74)
  Fatigue: Change at Day 841 (n=5) | 2.2 (21.37)
  Fatigue: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Fatigue: Change at Day 953 (n=1) | 66.7 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Fatigue: Change at Follow-up (n=12) | 5.6 (19.82)
  Nausea and vomiting: Baseline (n=52) | 4.8 (12.93)
  Nausea and vomiting: Change at Day 29 (n=47) | 1.4 (14.67)
  Nausea and vomiting: Change at Day 57 (n=45) | 4.1 (16.34)
  Nausea and vomiting: Change at Day 113 (n=41) | 10.2 (19.32)
  Nausea and vomiting: Change at Day 169 (n=32) | 1.0 (15.80)
  Nausea and vomiting: Change at Day 225 (n=28) | 1.2 (16.93)
  Nausea and vomiting: Change at Day 281 (n=23) | -0.7 (15.47)
  Nausea and vomiting: Change at Day 337 (n=14) | 1.2 (23.99)
  Nausea and vomiting: Change at Day 393 (n=19) | 1.8 (22.15)
  Nausea and vomiting: Change at Day 449 (n=17) | 5.9 (22.78)
  Nausea and vomiting: Change at Day 505 (n=20) | 1.7 (17.85)
  Nausea and vomiting: Change at Day 561 (n=17) | 4.9 (22.64)
  Nausea and vomiting: Change at Day 617 (n=14) | 11.9 (15.23)
  Nausea and vomiting: Change at Day 673 (n=11) | 6.1 (30.07)
  Nausea and vomiting: Change at Day 729 (n=11) | 0.0 (24.72)
  Nausea and vomiting: Change at Day 785 (n=10) | -1.7 (26.59)
  Nausea and vomiting: Change at Day 841 (n=5) | 6.7 (9.13)
  Nausea and vomiting: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Nausea and vomiting: Change at Day 953 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Nausea and vomiting: Change at follow-up (n=12) | 1.4 (11.14)
  Pain: Baseline (n=52) | 22.1 (23.04)
  Pain: Change at Day 29 (n=47) | 10.3 (22.40)
  Pain: Change at Day 57 (n=45) | 5.9 (26.39)
  Pain: Change at Day 113 (n=42) | 6.7 (25.25)
  Pain: Change at Day 169 (n=32) | 5.2 (29.77)
  Pain: Change at Day 225 (n=29) | 6.9 (35.50)
  Pain: Change at Day 281 (n=23) | 0.7 (34.26)
  Pain: Change at Day 337 (n=14) | -0.0 (26.95)
  Pain: Change at Day 393 (n=19) | -7.0 (27.95)
  Pain: Change at Day 449 (n=17) | -3.9 (27.97)
  Pain: Change at Day 505 (n=20) | 6.7 (32.17)
  Pain: Change at Day 561 (n=17) | 1.0 (32.53)
  Pain: Change at Day 617 (n=14) | 3.6 (25.47)
  Pain: Change at Day 673 (n=11) | -3.0 (37.87)
  Pain: Change at Day 729 (n=11) | -1.5 (32.88)
  Pain: Change at Day 785 (n=10) | 3.3 (33.15)
  Pain: Change at Day 841 (n=5) | -3.3 (24.72)
  Pain: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Pain: Change at Day 953 (n=1) | 33.3 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Pain: Change at follow-up (n=12) | 8.3 (33.71)
  Dyspnea: Baseline (n=52) | 18.6 (24.18)
  Dyspnea: Change at Day 29 (n=47) | -0.7 (23.56)
  Dyspnea: Change at Day 57 (n=45) | -0.7 (19.45)
  Dyspnea: Change at Day 113 (n=41) | -1.6 (18.18)
  Dyspnea: Change at Day 169 (n=32) | -3.1 (22.97)
  Dyspnea: Change at Day 225 (n=28) | 2.4 (29.99)
  Dyspnea: Change at Day 281 (n=23) | 0.0 (31.78)
  Dyspnea: Change at Day 337 (n=14) | -7.1 (32.50)
  Dyspnea: Change at Day 393 (n=19) | -5.3 (20.07)
  Dyspnea: Change at Day 449 (n=17) | -5.9 (24.25)
  Dyspnea: Change at Day 505 (n=20) | 1.7 (29.57)
  Dyspnea: Change at Day 561 (n=17) | 0.0 (26.35)
  Dyspnea: Change at Day 617 (n=14) | 4.8 (31.64)
  Dyspnea: Change at Day 673 (n=11) | -6.1 (32.72)
  Dyspnea: Change at Day 729 (n=11) | -3.0 (27.71)
  Dyspnea: Change at Day 785 (n=10) | 3.3 (24.60)
  Dyspnea: Change at Day 841 (n=5) | 0.0 (23.57)
  Dyspnea: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Dyspnea: Change at Day 953 (n=1) | 33.3 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Dyspnea: Change at follow-up (n=12) | -2.8 (22.29)
  Insomnia: Baseline (n=51) | 23.5 (30.03)
  Insomnia: Change at Day 29 (n=46) | -1.4 (30.60)
  Insomnia: Change at Day 57 (n=45) | -2.2 (30.48)
  Insomnia: Change at Day 113 (n=41) | -3.3 (28.68)
  Insomnia: Change at Day 169 (n=32) | -2.1 (31.61)
  Insomnia: Change at Day 225 (n=28) | -4.8 (38.18)
  Insomnia: Change at Day 281 (n=23) | 0.0 (36.24)
  Insomnia: Change at Day 337 (n=14) | -7.1 (37.39)
  Insomnia: Change at Day 393 (n=19) | -7.0 (36.14)
  Insomnia: Change at Day 449 (n=17) | -2.0 (32.21)
  Insomnia: Change at Day 505 (n=20) | -5.0 (31.11)
  Insomnia: Change at Day 561 (n=17) | -9.8 (36.83)
  Insomnia: Change at Day 617 (n=14) | -4.8 (34.24)
  Insomnia: Change at Day 673 (n=11) | -3.0 (43.34)
  Insomnia: Change at Day 729 (n=11) | -12.1 (34.23)
  Insomnia: Change at Day 785 (n=10) | -13.3 (39.13)
  Insomnia: Change at Day 841 (n=5) | -13.3 (50.55)
  Insomnia: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Insomnia: Change at Day 953 (n=1) | 33.3 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Insomnia: Change at follow-up (n=11) | -3.0 (23.35)
  Loss of appetite: Baseline (n=52) | 12.8 (25.70)
  Loss of appetite: Change at Day 29 (n=47) | 7.1 (31.80)
  Loss of appetite: Change at Day 57 (n=45) | 5.9 (33.55)
  Loss of appetite: Change at Day 113 (n=41) | 15.4 (34.24)
  Loss of appetite: Change at Day 169 (n=32) | 5.2 (35.02)
  Loss of appetite: Change at Day 225 (n=28) | 4.8 (38.18)
  Loss of appetite: Change at Day 281 (n=22) | 1.5 (31.67)
  Loss of appetite: Change at Day 337 (n=14) | -2.4 (42.29)
  Loss of appetite: Change at Day 393 (n=19) | 5.3 (35.60)
  Loss of appetite: Change at Day 449 (n=17) | 2.0 (36.27)
  Loss of appetite: Change at Day 505 (n=20) | -0.0 (34.20)
  Loss of appetite: Change at Day 561 (n=17) | 2.0 (36.27)
  Loss of appetite: Change at Day 617 (n=14) | 9.5 (20.37)
  Loss of appetite: Change at Day 673 (n=11) | -3.0 (43.34)
  Loss of appetite: Change at Day 729 (n=11) | -6.1 (35.96)
  Loss of appetite: Change at Day 785 (n=10) | -13.3 (42.16)
  Loss of appetite: Change at Day 841 (n=5) | 6.7 (43.46)
  Loss of appetite: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Loss of appetite: Change at Day 953 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Loss of appetite: Change at follow-up (n=12) | 8.3 (25.13)
  Constipation: Baseline (n=52) | 13.5 (22.15)
  Constipation: Change at Day 29 (n=47) | 5.0 (16.99)
  Constipation: Change at Day 57 (n=45) | 3.0 (17.15)
  Constipation: Change at Day 113 (n=41) | 4.1 (27.08)
  Constipation: Change at Day 169 (n=32) | 2.1 (28.00)
  Constipation: Change at Day 225 (n=28) | 0.0 (25.66)
  Constipation: Change at Day 281 (n=23) | 2.9 (22.28)
  Constipation: Change at Day 337 (n=14) | 4.8 (25.68)
  Constipation: Change at Day 393 (n=18) | -7.4 (21.56)
  Constipation: Change at Day 449 (n=17) | 0.0 (26.35)
  Constipation: Change at Day 505 (n=20) | 5.0 (29.17)
  Constipation: Change at Day 561 (n=17) | 0.0 (23.57)
  Constipation: Change at Day 617 (n=14) | -4.8 (17.82)
  Constipation: Change at Day 673 (n=11) | -6.1 (20.10)
  Constipation: Change at Day 729 (n=11) | -3.0 (10.05)
  Constipation: Change at Day 785 (n=10) | -3.3 (18.92)
  Constipation: Change at Day 841 (n=5) | -6.7 (14.91)
  Constipation: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Constipation: Change at Day 953 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Constipation: Change at follow-up (n=12) | 2.8 (22.29)
  Diarrhea: Baseline (n=52) | 8.3 (20.74)
  Diarrhea: Change at Day 29 (n=47) | 1.4 (16.96)
  Diarrhea: Change at Day 57 (n=45) | 5.9 (21.66)
  Diarrhea: Change at Day 113 (n=41) | 17.9 (28.96)
  Diarrhea: Change at Day 169 (n=32) | 16.7 (38.80)
  Diarrhea: Change at Day 225 (n=28) | 20.2 (26.20)
  Diarrhea: Change at Day 281 (n=23) | 29.0 (28.96)
  Diarrhea: Change at Day 337 (n=14) | 42.9 (33.15)
  Diarrhea: Change at Day 393 (n=19) | 33.3 (33.33)
  Diarrhea: Change at Day 449 (n=17) | 23.5 (25.72)
  Diarrhea: Change at Day 505 (n=20) | 35.0 (35.00)
  Diarrhea: Change at Day 561 (n=17) | 31.4 (27.56)
  Diarrhea: Change at Day 617 (n=14) | 40.5 (26.73)
  Diarrhea: Change at Day 673 (n=11) | 36.4 (37.87)
  Diarrhea: Change at Day 729 (n=11) | 27.3 (32.72)
  Diarrhea: Change at Day 785 (n=10) | 16.7 (17.57)
  Diarrhea: Change at Day 841 (n=5) | 20.0 (18.26)
  Diarrhea: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Diarrhea: Change at Day 953 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Diarrhea: Change at follow-up (n=12) | -11.1 (25.95)
  Financial difficulties: Baseline (n=51) | 15.0 (26.09)
  Financial difficulties: Change at Day 29 (n=45) | -3.0 (24.44)
  Financial difficulties: Change at Day 57 (n=33) | -8.1 (26.39)
  Financial difficulties: Change at Day 113 (n=41) | -5.7 (23.45)
  Financial difficulties: Change at Day 169 (n=32) | -3.1 (13.01)
  Financial difficulties: Change at Day 225 (n=28) | 1.2 (32.05)
  Financial difficulties: Change at Day 281 (n=23) | 1.4 (15.82)
  Financial difficulties: Change at Day 337 (n=14) | 0.0 (18.49)
  Financial difficulties: Change at Day 393 (n=19) | -1.8 (20.71)
  Financial difficulties: Change at Day 449 (n=16) | 2.1 (22.67)
  Financial difficulties: Change at Day 505 (n=19) | -1.8 (20.71)
  Financial difficulties: Change at Day 561 (n=17) | -2.0 (29.98)
  Financial difficulties: Change at Day 617 (n=14) | 0.0 (29.24)
  Financial difficulties: Change at Day 673 (n=11) | -6.1 (29.13)
  Financial difficulties: Change at Day 729 (n=11) | -6.1 (25.03)
  Financial difficulties: Change at Day 785 (n=10) | 10.0 (31.62)
  Financial difficulties: Change at Day 841 (n=4) | 8.3 (16.67)
  Financial difficulties: Change at Day 897 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Financial difficulties: Change at Day 953 (n=1) | 0.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Financial difficulties: Change at follow-up (n=12) | 0.0 (14.21)

6. Other Pre Specified Outcome: Population Pharmacokinetics of Axitinib (AG-013736)
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Day 1 (Pre-dose), Day 29, Day 57 and then every 8 weeks up to 139 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib
Serious Adverse Events (participants affected / at risk) | 28/52
Other Adverse Events (participants affected / at risk) | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=52)
Anaemia Not otherwise specified (NOS) (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia NOS (Cardiac disorders) | 3
Cardiomyopathy NOS (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericarditis NOS (Cardiac disorders) | 1
Diarrhoea NOS (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Weakness (General disorders) | 1
Bone infection NOS (Infections and infestations) | 1
Fungal infection NOS (Infections and infestations) | 1
Infusion site infection (Infections and infestations) | 1
Perianal abscess (Infections and infestations) | 1
Skin infection NOS (Infections and infestations) | 1
Blister (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Splenic haematoma (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in limb (Musculoskeletal and connective tissue disorders) | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spinal cord compression NOS (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Renal failure NOS (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hernia repair NOS (Surgical and medical procedures) | 1
Hypertension NOS (Vascular disorders) | 1
Hypertension aggravated (Vascular disorders) | 2
Hypotension NOS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=52)
Anaemia (Blood and lymphatic system disorders) | 7
Hypothyroidism (Endocrine disorders) | 4
Vision blurred (Eye disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 4
Anorectal discomfort (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 33
Dry mouth (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 11
Flatulence (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Haematochezia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 31
Proctalgia (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 4
Chest discomfort (General disorders) | 4
Chest pain (General disorders) | 7
Chills (General disorders) | 3
Fatigue (General disorders) | 33
Mucosal inflammation (General disorders) | 3
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 9
Bronchitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 11
Rhinitis (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 5
Tooth abscess (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 8
Weight decreased (Injury, poisoning and procedural complications) | 19
Decreased appetite (Metabolism and nutrition disorders) | 22
Dehydration (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 16
Hyperaesthesia (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 9
Peripheral sensory neuropathy (Nervous system disorders) | 4
Sensory disturbance (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 9
Haematuria (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 4
Erectile dysfunction (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Blister (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 18
Erythema (Skin and subcutaneous tissue disorders) | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 7
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 31
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.